CLINICAL TRIAL: NCT04188366
Title: Improving Family Engagement in First Episode Psychosis Care
Brief Title: Improving Family Engagement in Coordinated Specialty Care for First Episode Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Oladunni Oluwoye, Research Assistant Professor, Washington State University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17761-001; K01MH117457-01A1 (NIH)
Record Dates: First submitted 2019-11-27; First posted 2019-12-05 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Family Members
Keywords: Coordinated Specialty Care; Family Engagement; First Episode Psychosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAMES Modification (Experimental): 3-month trial of FAMES. Results from modifications will be used to by stakeholders (i.e., family members, client, providers, organizational leadership,) to inform finalization and implementation of FAMES
  Interventions: Behavioral: FAMES
- FAMES Pilot Trial (Experimental): Pilot testing of FAMES and implementation toolkit
  Interventions: Behavioral: FAMES; Behavioral: Treatment-as-Usual

INTERVENTIONS:
Behavioral: FAMES — Participants will receive three distinct and revolving components - early, continuous, and motivational contact - that incorporate motivational techniques and the Diagnostic and Statistical Manual of Mental Disorders 5TH Edition (DSM-5) Cultural Formulation Interview (CFI).
Behavioral: Treatment-as-Usual — Participants will receive usual services and family-based treatment offered
  Arms: FAMES Pilot Trial

SUMMARY:
Investigators aim to develop and evaluate a culturally informed family motivational engagement strategy (FAMES) and implementation toolkit for coordinated specialty care (CSC) programs for first episode psychosis. First, 5 family member participants will be recruited into a three-month trial of FAMES and implementation toolkit. The investigators will then conduct a 16-month non-randomized, stepped-wedge trial with 50 family members from 5 CSC programs in community-based mental health clinics.

DETAILED DESCRIPTION:
FAMES involves three distinct and revolving components - early, continuous, and motivational contact - that incorporate motivational techniques and the Diagnostic and Statistical Manual of Mental Disorders 5TH Edition (DSM-5) Cultural Formulation Interview (CFI).

The overarching objective of this study is to assess the feasibility and acceptability of a brief provider-led FAmily Engagement Motivational Strategy (FAMES) and its accompanying implementation toolkit. The investigators will also preliminary examine whether FAMES improves family engagement and retention in treatment, and motivation.

A total of 50 participants with a loved one enrolled in CSC program for FEP will be recruited from five CSC programs in Washington State to take part in a non-randomized stepped-wedge pilot trial. Each CSC program will represent a cluster and serve as its own control. A two-month implementation transition period will occur at each CSC program and during which providers will be introduced to the intervention using the implementation toolkits and trained to conduct FAMES. A 12-month open cohort design will be utilized to recruit approximately 50 family members during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older;
2. One family member (e.g., parent, guardian, aunt, uncle, spouse, grandparent, sibling, close friend) of an individual enrolled in a Washington State CSC program; and
3. Received no more than 6 months of services

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire-8 (CSQ-8) | Baseline through study completion, an average of 1 year; repeated measure to assess change through study completion
  Self-report measure to assess acceptability, a brief measure for family member participant. Items are scored from 1 to 4. Possible total scores range from 8 to 32, with higher scores (>23) indicating greater satisfaction.
Youth Services Survey-Families (YSS-F) | Baseline through study completion, an average of 1 year; repeated measure to assess change through study completion
  Self-report measure to assess acceptability in the following domains: appropriateness, participation, cultural sensitivity, social connectedness, and outcomes. Items in a domain are summed and divided by the total number of items, and scores greater than 3.5 are reported in the positive range for the domain.
Qualitative interviews | Month 1 of treatment period and month 1 follow-up period; repeated measure to assess change in acceptability and feasibility
  Interviews with providers and family member participants to assess acceptability and of FAMES

SECONDARY OUTCOMES:
Level of Engagement to measure effectiveness of FAMES | Baseline through study completion, an average of 1 year; repeated measure to assess change through study completion
  Provider reported service utilization. Total number of contact hours between provider and family member to measure engagement
Rate of Retention to measure effectiveness of FAMES | Baseline through study completion, an average of 1 year; repeated measure to assess change through study completion
  Provider reported service utilization. Percentage of families that dropout (family member declined or missed three consecutive appointments).
Burden Assessment Scale (BAS) | Baseline through study completion, an average of 1 year; repeated measure to assess change through study completion
  Self-report measure to assess family functioning. Total possible scores range from 10 to 171 (higher scores indicating greater burden)
Iowa Cultural Understanding Assessment | Baseline through study completion, an average of 1 year; repeated measure to assess change through study completion
  Self-report measure to assess provider cultural competence. All items are scored from 1=strongly disagree to 5=strongly agree. Total scores range from 25 to 125 (higher scores indicating great cultural competence)
Treatment Self-Regulation Questionnaire (TSRQ) | Baseline through study completion, an average of 1 year; repeated measure to assess change through study completion
  Self-report measure to assess motivation. Scale ranges from 1=not at all true to 7=very true.

OTHER OUTCOMES:
Organizational Readiness to Change Assessment (ORCA) | Baseline through study completion, an average of 1 year; repeated measure to assess change through study completion
  Self-report provider measure to assess assess evidence assessment, contextual readiness and facilitation needs. All items are scored from 1=strongly disagree to 5=strongly agree

CONTACTS AND LOCATIONS:
Locations (1):
- New Journeys: Coordinated specialty care, Yakima, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oluwoye O, Dyck D, McPherson SM, Lewis-Fernandez R, Compton MT, McDonell MG, Cabassa LJ. Developing and implementing a culturally informed FAmily Motivational Engagement Strategy (FAMES) to increase family engagement in first episode psychosis programs: mixed methods pilot study protocol. BMJ Open. 2020 Aug 26;10(8):e036907. doi: 10.1136/bmjopen-2020-036907. PMID 32847910